CLINICAL TRIAL: NCT01798966
Title: The Effects of Orbital Decompression Surgery on Intraocular Pressure Patterns in Patient With Thyroid Eye Disease Undergoing 24 Hour Continuous IOP Monitoring With the SENSIMED Triggerfish®
Brief Title: Twenty-four Hour Intraocular Pressure Patterns in Patients With Uncontrolled Thyroid Eye Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sensimed AG (Industry)
Collaborators: University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TF-1111
Record Dates: First submitted 2013-02-21; First posted 2013-02-26 (Estimated); Results first posted 2015-03-02 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-02

CONDITIONS: Thyroid Eye Disease
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SENSIMED Triggerfish (Experimental): Sensimed Triggerfish device will be worn by each subject for 24h
  Interventions: Device: SENSIMED Triggerfish

INTERVENTIONS:
Device: SENSIMED Triggerfish
  Other Names: Contact lens sensor intented to continuously record IOP pattern for up to 24 hours

SUMMARY:
Patients with Thyroid Eye Disease (TED) often have enlarged extraocular muscles and higher orbital fat contents due to their disease process. The confined space of the orbit cannot hold the enlarged orbital contents creating a forward displacement and/or compression of the globe with a rise in intraocular pressure (IOP). Many of these patients undergo surgical decompression, a procedure that fractures orbital bones, in order to allow more space for the enlarged orbital contents to occupy. To date, there is no data that shows intraocular patterns over a 24-hour period in patients with mechanical compression on the globe as in TED. It is not know if the pattern of IOP is more consistent with normal IOP patterns, glaucomatous patterns, or perhaps completely different then either. The goal of this project is to investigate patterns of IOP in patients requiring orbital decompression because of orbital congestion. Changes in IOP during a 24-hour period will be studied with a contact-lens embedded sensor that provides continuous data. This device has previously been investigated and shown to be safe and well-tolerated. Monitoring the pattern in these patients will allow us to compare Thyroid TED patterns of IOP with those of normal and glaucomatous patients. Also, testing these patients before and after orbital decompression surgery will allow characterization of how intraocular pressure changes once the mechanical compression on the globe is relieved.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to comply with the study procedures
* 18-80 years old
* Subjects diagnosed with Thyroid Eye Disease based on both endocrinology studies showing autoimmune dysfunction consistent with Graves' Disease as well as orbital imaging studies manifesting characteristics consistent with Thyroid Eye Disease.
* Ability to understand the character and individual consequences of the study
* Subject has consented to be in the trial

Exclusion Criteria:

* Subjects with contraindications for wearing contact lenses
* Severe ocular surface disease
* Keratoconus or other corneal abnormality
* Severe ocular inflammation
* Full frame metal glasses during SENSIMED Triggerfish® monitoring
* Known hypersensitivity to silicone, plaster or ocular anesthesia (proparacaine)
* Simultaneous participation in other clinical studies
* Diagnosis of glaucoma

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald O Kikkawa, MD, Principal Investigator — University of California, San Diego
Locations (1):
- Shiley Eye Center, University of California, San Diego, La Jolla, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- SENSIMED Triggerfish: All patients included in the device group
Period: Overall Study
Arm/Group | SENSIMED Triggerfish
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SENSIMED Triggerfish
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (21.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 10
Tolerability of CLS [Mean (Standard Deviation); unit: units on a scale] — Subjective comfort level using a number between 0-10 with values ranging from 0 (no discomfort) to 10 (very severe discomfort)
  units on a scale | 1.5 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in IOP Before and After Orbital Decompression Surgery
Description: To investigate the difference in SENSIMED Triggerfish output during transition from wake to sleep states before and after orbital decompression
Time Frame: 24 hours
Measure: Median (Standard Deviation); unit: mVEq (Sensismed Triggerfish output unit)
Groups:
- SENSIMED Triggerfish: SENSIMED Triggerfish worn for 24h
Arm/Group | SENSIMED Triggerfish
Number analyzed (Participants) | 10
mVEq (Sensismed Triggerfish output unit) | 18 (43.8)

2. Secondary Outcome: IOP Patterns
Description: The pattern of IOP in patients with TED will be compared with the pattern of IOP readings in normal subjects as well as glaucomatous patients
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: mvEq
Arm/Group | SENSIMED Triggerfish
Number analyzed (Participants) | 10
mvEq | 102.2 (52.6)

3. Other Pre Specified Outcome: Adverse Events and Serious Adverse Events
Description: Safety will be evaluated throughout the duration of the study by collecting all adverse events
Time Frame: 4 days
Measure: Number; unit: Number of AE
Arm/Group | SENSIMED Triggerfish
Number analyzed (Participants) | 10
Number of AE | 3

ADVERSE EVENTS:
Time Frame: From inform consent signature to 30 days after last exposure to device
Arm/Group | SENSIMED Triggerfish
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SENSIMED Triggerfish (N=10)
Mild blurred vision (Eye disorders) | 5
Mild hyperemia and palpebral conjunctiva (Eye disorders) | 10
Superficial Punctate keratitis (Eye disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No